CLINICAL TRIAL: NCT07126067
Title: Effect of Dynamic Compliance and Individualized PEEP Value Based on Lung Ultrasound on Postoperative Diaphragmatic Function in Pediatric Patients Undergoing Laparoscopic Abdominal Surgery
Brief Title: Postoperative Diaphragm Function in Pediatric Laparoscopic Abdominal Surgery Using Compliance and PEEP Guided by Lung Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Yasin Tire, MD, Anesthesiologist, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Study Pedpeep
Record Dates: First submitted 2025-03-02; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: PEEP by Lung Ultrasound; PEEP With Dynamic Compliance
Keywords: PEEP; Lung Ulrasound; Laparoscopic surgery; Pediatric patients.

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients who underwent individualized PEEP with lung USG (Active Comparator): In participants from Group U, PEEP will initially be set at 5 cmH2O and adjusted based on lung ultrasound (USG) findings. If the lung consolidation score is ≥ 2, the PEEP level will be incrementally increased by 2 cmH2O, with USG reassessments every 5 minutes, until a score < 2 is achieved. This process will be repeated after pneumoperitoneum, peritoneal deflation, and positional changes during surgery to establish an individualized PEEP level. The maximum PEEP value is limited to 20 cmH2O, with a plateau pressure (Pplat) cap of 30 cmH2O and a peak inspiratory pressure (PIP) limit of 40 cmH2O.
  Interventions: Procedure: Lung Ultrasound and PEEP Application
- Application of PEEP with Dynamic Compliance (Active Comparator): PEEP starts at 5 cmH2O after endotracheal intubation. The ventilator (Mindray) will automatically monitor dynamic compliance (TV/Ppeak-PEEP) 5 minutes after endotracheal insertion. PEEP will rise 3 cmH2O. The Cdyn value will be tested again after six breathing cycles, and if it increases, PEEP will be increased by 2 cmH2O. If Cdyn readings decrease during six consecutive automatic measurements, the participant's optimal PEEP level will be the prior measurement's PEEP.
  To calculate Cdyn-based PEEP, the same technique will be repeated following pneumoperitoneum, peritoneal deflation, and positional changes during operation.
  For dynamic compliance-based PEEP participants (Group D), the maximum PEEP value will be 20 cmH2O, the plateau pressure (Pplat) limit 30 cmH2O, and the peak inspiratory pressure (PIP) limit 40 cmH2O.
  Interventions: Procedure: Application of PEEP with Dynamic Compliance
- Control Group (No Intervention): Control group participants will receive conventional mechanical ventilation without PEEP modification interventions. PEEP shall stay at 5 cmH2O during surgery unless clinically indicated to change (e.g., substantial hypoxaemia or haemodynamic instability).
  These subjects will not undergo Cdyn or LUS measures. Instead, institutional protocols will guide intraoperative monitoring and treatment. Depending on clinical measures like oxygen saturation (SpO2), end-tidal carbon dioxide (EtCO2), and arterial blood gas (ABG), the anaesthesiologist may adjust ventilator settings.
  The control group serves as a baseline for comparison with the intervention groups (LUS or Cdyn-based PEEP adjustments) to determine if individualised PEEP techniques improve clinical results.

INTERVENTIONS:
Procedure: Lung Ultrasound and PEEP Application — Application of Lung Ultrasound and PEEP After intubation, PEEP starts at 5 cmH2O. The first lung ultrasound (USG) is performed after 5 minutes. If the lung consolidation score is ≥2, PEEP increases by 2 cmH2O and is reassessed every 5 minutes until the score is <2. If <2, PEEP remains unchanged as the optimal level. This process is repeated after pneumoperitoneum, peritoneal deflation, and position changes. In Group U, PEEP is determined by USG, with a maximum of 20 cmH2O, a plateau pressure of 30 cmH2O, and a peak inspiratory pressure of 40 cmH2O.
  Arms: Patients who underwent individualized PEEP with lung USG
Procedure: Application of PEEP with Dynamic Compliance — Application of PEEP with Dynamic Compliance
  * After endotracheal intubation, PEEP will be applied as 5 cmH2O.
  * The first dynamic compliance (TV/Ppeak-PEEP) monitoring will be performed automatically by the ventilator (Mindray) 5 minutes after endotracheal intubation, and the PEEP value will be increased by 3 cmH2O. The obtained Cdyn value will be repeated after six respiratory cycles, and if there is an increase, the PEEP value will be increased by 2 cmH2O. When a decreasing trend is observed in the Cdyn value as a result of consecutive automatic measurements of 6 respiratory cycles, the PEEP value applied in the previous measurement will be determined as the most appropriate PEEP value for the participant.
  Arms: Application of PEEP with Dynamic Compliance

SUMMARY:
Protective ventilation strategies and alveolar recruitment maneuvers (ARM) are employed in patients with acute lung injury (ALI) and acute respiratory distress syndrome (ARDS) to improve oxygenation, prevent alveolar collapse, and reduce ventilation-induced lung injury. Recruitment maneuvers aim to open and maintain alveoli. While positive effects on oxygenation have been observed in adults, limited data in children make the clinical efficacy of these strategies uncertain. Careful application and the development of individualized treatment protocols are recommended.

DETAILED DESCRIPTION:
Experimental studies have proven a relationship between inappropriate ventilation measures and delayed or even worsened recovery from acute pulmonary injury. Therefore, the importance of protective ventilation combined with recruitment maneuvers emerges. In clinical practice, this relationship is believed to significantly reduce morbidity, mortality, and injuries caused by mechanical ventilation.

It is indicated in patients with severe hypoxemia, often due to acute lung injury caused by pneumonia or sepsis. The main contraindications are hemodynamic instability, pneumothorax, and intracranial hypertension. Experimental studies have shown that lung-protective ventilation has beneficial effects on both oxygenation and alveolar collapse. In children, lung-protective ventilation leads to significant reductions in alveolar collapse, lower oxygen requirements, improved pulmonary compliance, and decreased bronchopulmonary dysplasia. However, studies conducted on children are limited.

Recent changes have been made regarding how children with acute hypoxemic respiratory failure are ventilated. Lachmann proposed the "open lung concept," which involves opening the lungs and keeping them open during mechanical ventilation. ARM has been used for over two decades in mechanically ventilated patients with severe lung injury. Its most significant physiological outcome is the improvement in oxygenation in patients with lung damage. The procedure is typically followed by adjustments in PEEP levels, which play a fundamental role in maintaining the effectiveness of ARM. ARM is also used to prevent alveolar collapse during low tidal volume mechanical ventilation. However, its primary purpose is to protect the lungs from ventilator-induced injuries. PEEP has a key role in preventing atelectrauma and maintaining the maneuver's effectiveness. In clinical practice, these strategies are believed to significantly reduce morbidity and mortality.

In this study, it is aimed to define the limits of "diaphragm-protective ventilation" based on the clinical outcomes of our patients by evaluating the effects of different PEEP levels adjusted during laparoscopic abdominal surgery in pediatric patients. Additionally, it will be seeked to assess the impact of positive end-expiratory pressure levels on diaphragm thickness.

Our primary hypothesis is that, in patients where ideal PEEP is applied based on dynamic compliance measured with ultrasound (USG), diaphragm values will return closer to baseline values compared to those where recruitment maneuvers and ideal PEEP are applied.

Secondly, it is aimed to investigate the effects of calculating ideal PEEP using dynamic compliance measured with USG on hospital length of stay, intraoperative hemodynamic parameters, and respiratory parameters.

ELIGIBILITY:
Inclusion Criteria:

* Participants meeting the following criteria will be included in the study:
* Aged 7 to 12 years
* ASA classification I, II, or III
* Undergoing elective laparoscopic abdominal surgery

Exclusion Criteria:

Participants with any of the following conditions will be excluded from the study:

* Age <7 or >12 years
* ASA classification > III
* Uncontrolled bronchial asthma
* Presence of bullous lung disease
* Decompensated heart failure (NYHA Stage III-IV)
* History of lung surgery
* Increased intracranial or intraocular pressure
* Advanced hepatic or renal failure
* Parental refusal to participate in the study

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2024-12-25 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Diaphragm thickness 1 | Baseline measurement prior to anesthesia induction (within 30 minutes before surgery).
  Diaphragm Thickness Measurement In the supine position, diaphragm thickness will be measured at the junction of the midaxillary line, between the 8th or 9th intercostal spaces on the right side. Using a high-frequency linear probe and ultrasound (DC-60 Diagnostic Ultrasound, Shenzhen Mindray, China), measurements will be recorded during inspiration and expiration. Once a clear diaphragm image is obtained, the skin at the probe's caudal end will be marked with indelible ink. All images will be captured with the probe in the same position. The average of inspiratory and expiratory diaphragm thickness will be used to calculate the diaphragm thickness ratio.
Diaphragm thickness 2 | Immediately after extubation in the operating room (within 5 minutes of extubation).
  Diaphragm Thickness Measurement In the supine position, diaphragm thickness will be measured at the junction of the midaxillary line, between the 8th or 9th intercostal spaces on the right side. Using a high-frequency linear probe and ultrasound (DC-60 Diagnostic Ultrasound, Shenzhen Mindray, China), measurements will be recorded during inspiration and expiration. Once a clear diaphragm image is obtained, the skin at the probe's caudal end will be marked with indelible ink. All images will be captured with the probe in the same position. The average of inspiratory and expiratory diaphragm thickness will be used to calculate the diaphragm thickness ratio.
Diaphragm thickness 3 | 30 minutes after surgery completion (within the postoperative recovery period, up to 30 minutes).
  Diaphragm Thickness Measurement In the supine position, diaphragm thickness will be measured at the junction of the midaxillary line, between the 8th or 9th intercostal spaces on the right side. Using a high-frequency linear probe and ultrasound (DC-60 Diagnostic Ultrasound, Shenzhen Mindray, China), measurements will be recorded during inspiration and expiration. Once a clear diaphragm image is obtained, the skin at the probe's caudal end will be marked with indelible ink. All images will be captured with the probe in the same position. The average of inspiratory and expiratory diaphragm thickness will be used to calculate the diaphragm thickness ratio.

SECONDARY OUTCOMES:
Definition and Assessment of Postoperative Pulmonary Complications (PPCs) | From the end of surgery until 24 hours postoperatively.
  Definition and Assessment of Postoperative Pulmonary Complications (PPCs)
  PPCs will be considered positive if at least one of the following conditions occurs within the first 24 hours postoperatively:
  Mild Respiratory Failure: PaO₂ < 60 mmHg or SpO₂ < 90% requiring ≤2 L/min O₂ therapy.
  Moderate Respiratory Failure: PaO₂ < 60 mmHg or SpO₂ < 90% requiring >2 L/min O₂ therapy.
  Severe Respiratory Failure: Need for non-invasive or invasive ventilation. ARDS: Defined by the Berlin criteria. Bronchospasm: Newly detected expiratory wheezing treated with bronchodilators. Pulmonary Infection Pleural Effusion Pulmonary Atelectasis Cardiopulmonary Edema Pneumothorax

CONTACTS AND LOCATIONS:
Locations (1):
- Yasin Tire, Konya, Meram, Turkey (Türkiye)